CLINICAL TRIAL: NCT05367531
Title: Quantitative Assessment of Injectable Medication Delivery Practices
Brief Title: Assessment of Injectable Medication Platforms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Canadian Forces Health Services Centre Ottawa (Other)
Responsible Party: Principal Investigator, Gaurav Gupta, Principal Investigator, Canadian Forces Health Services Centre Ottawa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020-046
Record Dates: First submitted 2022-04-28; First posted 2022-05-10 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Overdose Antidote; Bleeding; Allergic Reaction
Keywords: autoinjector; needle; syringe; medication
MeSH Terms: conditions — Hemorrhage; Hypersensitivity

STUDY DESIGN:
Intervention Model Description: For each scenario participants will be asked to administer/inject the "medication" (likely saline or air) using various methods: 1) standard protocol , 2) Autoinjector 3) Pre-filled syringes. For each scenario the appropriate medication administration type will have to be selected amongst groups of options: 1) autoinjectors equivalents (ie medication, needle and syringe attached) 2) prefilled syringes where a needle is attached prior to administration; and 3) standard protocol (i.e. drawing medication from the vial and injecting via syringe/22 gauge needle). Medications options will include 1) Naloxone (opioid overdose) 2) Epinephrine (anaphylaxis) 3) Tranexamic acid (bleeding).
Masking Description: The order of administration for each scenario and injection type will be randomized to exclude any bias. To minimize risk to participants, active drug products and live/loaded autoinjectors will not be used. The target injection will be placed in an inanimate object (e.g. orange) or phantom simulator (i.e. inanimate object such as a gel or organic material such as jello or fruit to simulate an injection experience).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Injection Scenario (Experimental): For each scenario participants will be asked to administer/inject the "medication" (likely saline or air) using various methods: 1) standard protocol , 2) Autoinjector 3) Pre-filled syringes. For each scenario the appropriate medication administration type will have to be selected amongst groups of options: 1) autoinjectors equivalents (ie medication, needle and syringe attached) 2) prefilled syringes where a needle is attached prior to administration; and 3) standard protocol (i.e. drawing medication from the vial and injecting via syringe/22 gauge needle). Medications options will include 1) Naloxone (opioid overdose) 2) Epinephrine (anaphylaxis) 3) Tranexamic acid (bleeding).
  Interventions: Device: Autoinjector; Device: Standard Injector; Device: Prefilled

INTERVENTIONS:
Device: Autoinjector — For each scenario the appropriate medication administration type will have to be selected amongst groups of options: 1) autoinjectors equivalents (ie medication, needle and syringe attached) 2) prefilled syringes where a needle is attached prior to administration; and 3) standard protocol (i.e. drawing medication from the vial and injecting via syringe/22 gauge needle). Medications options will include 1) Naloxone (opioid overdose) 2) Epinephrine (anaphylaxis) 3) Tranexamic acid (bleeding).
  The order of administration for each scenario and injection type will be randomized to exclude any bias. To minimize risk to participants, active drug products and live/loaded autoinjectors will not be used. The target injection will be placed in an inanimate object (e.g. orange) or phantom simulator (i.e. inanimate object such as a gel or organic material such as jello or fruit to simulate an injection experience).
Device: Standard Injector — For each scenario the appropriate medication administration type will have to be selected amongst groups of options: 1) autoinjectors equivalents (ie medication, needle and syringe attached) 2) prefilled syringes where a needle is attached prior to administration; and 3) standard protocol (i.e. drawing medication from the vial and injecting via syringe/22 gauge needle). Medications options will include 1) Naloxone (opioid overdose) 2) Epinephrine (anaphylaxis) 3) Tranexamic acid (bleeding).
  The order of administration for each scenario and injection type will be randomized to exclude any bias. To minimize risk to participants, active drug products and live/loaded autoinjectors will not be used. The target injection will be placed in an inanimate object (e.g. orange) or phantom simulator (i.e. inanimate object such as a gel or organic material such as jello or fruit to simulate an injection experience).
Device: Prefilled — For each scenario the appropriate medication administration type will have to be selected amongst groups of options: 1) autoinjectors equivalents (ie medication, needle and syringe attached) 2) prefilled syringes where a needle is attached prior to administration; and 3) standard protocol (i.e. drawing medication from the vial and injecting via syringe/22 gauge needle). Medications options will include 1) Naloxone (opioid overdose) 2) Epinephrine (anaphylaxis) 3) Tranexamic acid (bleeding).
  The order of administration for each scenario and injection type will be randomized to exclude any bias. To minimize risk to participants, active drug products and live/loaded autoinjectors will not be used. The target injection will be placed in an inanimate object (e.g. orange) or phantom simulator (i.e. inanimate object such as a gel or organic material such as jello or fruit to simulate an injection experience).

SUMMARY:
Background:

While medical advances for in-hospital care rapidly evolve, a mainstay of effective pre-hospital care remains the ability to treat medical emergencies such as anaphylaxis, prolonged seizure, overdose, or uncontrolled bleeding, through rapid administration of appropriate medication. Autoinjectors are used globally to deliver medications in a timely manner, often in environments where immediate access to medical facilities is limited. Rapid administration of intramuscular medication delivery is essential where oral or intravenous delivery is either not possible or ineffective. The purpose of the proposed study seeks to determine the efficiency various types of medication injection administration.

DETAILED DESCRIPTION:
Research Objective:

To understand the efficiency of injectable medication delivery in the Canadian Forces and civilian world for improved care delivery in military and pre-hospital environments.

Participants:

Approximately thirty (30) participants will be recruited for the study.

Methods:

Data will be obtained on the technical comparison of efficiency for pre-filled syringes to the current standards of administration. The timing and accuracy for administering saline to an inanimate object using the traditional methods versus a pre-filled medication syringes will be compared.

Risks and Risk Mitigation:

The participants in this study are all practicing military personnel who are able to give free and informed consent. To reduce undue influence, LCol Meredith and Dr Gupta will not be involved in recruitment. As a result, these participants are a low vulnerability group. The risk of any adverse events is low since data scenarios, and participants may choose to skip any questions or scenarios that participants do not wish to do. Investigators will remind all participants that their participation is voluntary, and that they may choose to withdraw or stop at any time.

Benefits and Military Significance:

The proposed study will be the first of its kind to assess the efficiency of various injectable medication delivery platforms. This data will provide a background for improving injectable drug delivery practices in various setting (eg military and pre-hospital settings), including the potential to inform novel medical device development.

ELIGIBILITY:
Inclusion Criteria:

* any participant over the age of 18 able to provide consent

Exclusion Criteria:

* only participants with pre specified conditions impacting cognitive and/or manual dexterity will be excluded
* recent substance use
* non health care workers injection with experience with medication injection in last 12 months

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-04-30 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in medication Injection/delivery time for each trial | immediately after intervention
  Time in seconds will be measured from the start of the scenario and stopped once the medication has been delivered to the orange.

SECONDARY OUTCOMES:
Number of injection failures and/or injuries associated with each trial | immediately after intervention
  Any human errors or device failures will be recorded
Perceived difficulty of injection based on type of system | immediately after intervention
  On a scale of 1-5 participants will rate difficult using autoinjector, prefilled and standard medication delivery systems. Going from 1-5 represents a decreasing degree of difficulty (hardest =5 and easiest = 1 with 3 being neutral)

CONTACTS AND LOCATIONS:
Overall Officials: Gaurav Gupta, MD, Principal Investigator — CAF
Locations (1):
- Canadian Forces, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No